CLINICAL TRIAL: NCT03287258
Title: Digital Perineal Massage and Pelvic Floor Muscle Exercise as an Antenatal Program for Prevention of Perineal Trauma in Elderly Women, a Randomized Controlled Trial.
Brief Title: Perineal Preparation for Pregnant Ladies.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amira S Dieb, Department of Obstetrics and Gynecology, Kasr Al-Ainy hospital, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: perineal preparation study
Record Dates: First submitted 2017-07-22; First posted 2017-09-19 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Delivery; Trauma; Pelvic Floor; Perineal Rupture, Obstetric; Pelvic Floor Muscle Weakness
Keywords: perineal massage; health education; perineal tear; episiotomy; pelvic floor muscle exercise
MeSH Terms: conditions — Wounds and Injuries; Health Education

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three program (Active Comparator): 200 patients are subjected to educational Pelvic floor dysfunction prevention program with perineal massage and Pelvic floor muscle exercise.
  Interventions: Other: 3 program
- one program (Active Comparator): 200 patients are subjected to educational Pelvic floor dysfunction prevention program
  Interventions: Other: one program

INTERVENTIONS:
Other: 3 program — The participants will receive 3 programs.The educational pelvic floor dysfunction prevention program, pelvic floor muscle exercise program and perineal massage program will be educated by an investigator during the participant visit 4 weeks before her due date
  Arms: three program
Other: one program — The participants will receive one program. That is the educational pelvic floor dysfunction prevention program.The instructions of the program will be given by an investigator once during the participant visit 4 weeks before her due date.
  Arms: one program

SUMMARY:
Pregnant participants will be recruited at the obstetrics outpatient clinic during their visits 4 weeks before the due date. They are randomized into two groups. The first group will be educated to do digital perineal massage. They will be also educated to do pelvic floor muscle exercises and will receive the usual education program for strengthening the pelvic floor. The second group will receive the usual education program for strengthening the pelvic floor. Occurrence of perineal laceration will be reported at time of delivery.

DETAILED DESCRIPTION:
Pregnant participants will be recruited at the obstetrics outpatient clinic during their visits 4 weeks before the due date. They are randomized into two groups. The first group will be educated to do digital perineal massage. They will be also educated to do pelvic floor muscle exercises and will receive the usual educational pelvic floor dysfunction prevention program for strengthening the pelvic floor. The second group will receive the usual education program for strengthening the pelvic floor. Occurrence of perineal laceration will be reported at time of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 35 years old
* Primigravida or multi gravida

Exclusion Criteria:

* History of chronic constipation
* History of chronic cough
* Current or past urinary or anal incontinence
* History of genital prolapse before pregnancy
* History of neuromuscular disorders or connective tissue disorders
* History of medical disorders
* History of preterm or precipitate labour
* History of premature preterm rupture of membranes.
* Genital infections

Ages: 35 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
perineal tears Proportion of perineal tears will be assessed by an investigator who will attend the participant delivery | At 15 minutes from delivery
  Proportion of participants who have perineal tears

SECONDARY OUTCOMES:
episiotomy need Proportion of participants who need episiotomy at time of delivery will be assessed by an investigator | At 15 minutes from delivery
  Proportion of participants who need episiotomy at time of delivery
Duration of the second stage of labour | 2 hours
  Duration of the second stage of labour will be assessed by an investigator

CONTACTS AND LOCATIONS:
Overall Officials: Amira Dieb, MD, Principal Investigator — KasrAlainiH
Locations (1):
- KasralainiH, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No